CLINICAL TRIAL: NCT01023659
Title: An Innovative Approach to Maximizing the Impact of Efficacious Pharmacotherapies on Smoking Cessation Attempts.
Brief Title: Distribution of Bupropion and Varenicline to Increase Smoking Cessation Attempts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Dr. Peter Selby, Clinical Director, Addictions Program, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 068/2009
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Tobacco Use Disorder; Smoking; Smoking Cessation
Keywords: Smoking cessation; Bupropion; Varenicline; Population-level; Mass distribution; Drug Therapy
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Bupropion; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bupropion + motivational emails (Active Comparator): participants receive Zyban (300mg/day) plus weekly motivational emails for 12 weeks.
  Interventions: Drug: bupropion; Behavioral: motivational emails
- Varenicline + motivational emails (Active Comparator): participants receive Champix (2mg/day) plus weekly motivational emails for 12 weeks.
  Interventions: Drug: varenicline; Behavioral: motivational emails
- Motivational emails (Active Comparator): participants receive weekly motivational emails for 12 weeks.
  Interventions: Behavioral: motivational emails

INTERVENTIONS:
Drug: bupropion — bupropion, 150 mg twice daily plus weekly motivational emails for 12 weeks
  Other Names: Zyban
  Arms: Bupropion + motivational emails
Drug: varenicline — varenicline, 1 mg twice daily plus weekly motivational emails for 12 weeks
  Other Names: Champix
  Arms: Varenicline + motivational emails
Behavioral: motivational emails — brief motivational emails, sent weekly for 12 weeks

SUMMARY:
Bupropion and varenicline are indicated for smoking cessation. The objectives of this study are two-fold: (1) to explore the logistic feasibility of distributing bupropion and varenicline free of charge to treatment-seeking smokers in the province of Ontario, Canada and (2) to evaluate the real-world effectiveness of bupropion and varenicline treatment in Ontario compared to a no-drug comparison group. In an open label study, Ontario smokers who smoke 10 or more cigarettes per day and intend to quit smoking in the next 30 days, will enroll via the study website, visit their physician to receive a prescription for bupropion or varenicline for 12 weeks or neither if they so choose, forming the no-drug comparison group. All participants will receive weekly motivational emails for 12 weeks. Abstinence measures will be taken at 4, 8 and 12 weeks and at 6 and 12 months. The proportion of eligible participants who were able to confirm an appointment with a physician to receive the prescription will be also measured.

DETAILED DESCRIPTION:
Bupropion and varenicline are effective pharmacotherapies for smoking cessation, but their population level impact is limited by a combination of factors. Both bupropion and varenicline are only available through prescription, however smoking cessation clinics are few in number and only about 25% of smokers receive information on smoking cessation aids from their healthcare provider. Mass distribution approaches, bypassing clinics and physicians, have been successful for nicotine replacement therapy in many jurisdictions, including Ontario. However, bupropion and varenicline have the potential to make a greater impact given their superior results from the clinical trials. Bupropion and varenicline present a unique challenge as they are prescribed medications, therefore we have proposed a variant of the mass distribution method to test whether it is practical to distribute them to a large number of people over a expansive geographic area (i.e., Ontario).

We hypothesize that engaging smokers with the opportunity to receive free bupropion or varenicline, to initiate an appointment with their physician to obtain a prescription that would be filled and mailed to the smoker from a central pharmacy would be a logistically feasible approach to reach high number of smokers from a wide geographic area. Our second hypothesis is that consistent with the results from clinical studies, in the general population varenicline would be associated with a higher abstinence rate than bupropion, and both varenicline and bupropion groups would achieve higher abstinence rates than those making quit attempts without any pharmacotherapy aid.

This is an open label, proof-of-concept study, wherein 2000 eligible participants will have the opportunity to receive bupropion (Zyban®) or varenicline (Champix®) for 12 weeks in conjunction with weekly motivational emails. Eligible participants will discuss with their doctor which of the two medications is appropriate for them to use as smoking cessation aid. It is also possible that the participant and his/her doctor may decide not to pursue smoking cessation using either of these medications. These participants will form a third intervention group, receiving only the weekly motivational emails. All participants will set a quit date of their choosing, but those receiving medication will set a quit date 7 days after starting the medication. The participants will enroll in the study via the study's website, at which time they will read the consent form, answer the eligibility questions and complete the baseline questionnaire. Data related to the outcome measures and adverse events will be collected at 4, 8 and 12 weeks after the start of treatment and at 6 and 12 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female, at least 18 years of age, resident of Ontario, smoke at least 10 cigarettes per day, had smoked daily for at least the past 3 months, had smoked at least 100 cigarettes in their lifetime and intended to quit smoking in the next 30 days.

Exclusion Criteria:

* history of brain injury or seizure(s); pregnancy, lactation or risk of becoming pregnant; allergy or sensitivity to bupropion or varenicline; current use of monoamine oxidase inhibitors (MAOIs), thioridazine, varenicline or buproprion; severe liver impairment; or history of anorexia and /or bulimina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 893 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MD, MHSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Selby P, Hussain S, Voci S, Zawertailo L. Empowering smokers with a web-assisted tobacco intervention to use prescription smoking cessation medications: a feasibility trial. Implement Sci. 2015 Oct 1;10:139. doi: 10.1186/s13012-015-0329-7. PMID 26429100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants visited the study website, provided consent and completed an on-line assessment. Eligible participants received a personalized script to take to their physician, who could prescribe varenicline or bupropion for 12 weeks, or neither.
Groups:
- Bupropion + Motivational Emails: participants receive Zyban (300mg/day) plus weekly motivational emails for 12 weeks.
  bupropion : bupropion, 150 mg twice daily plus weekly motivational emails for 12 weeks
  motivational emails : brief motivational emails, sent weekly for 12 weeks
- Motivational Emails: participants receive weekly motivational emails for 12 weeks.
  motivational emails : brief motivational emails, sent weekly for 12 weeks
- Varenicline + Motivational Emails: participants receive Champix (2mg/day) plus weekly motivational emails for 12 weeks.
  motivational emails : brief motivational emails, sent weekly for 12 weeks
  varenicline : varenicline, 1 mg twice daily plus weekly motivational emails for 12 weeks
Period: Overall Study
Arm/Group | Bupropion + Motivational Emails | Motivational Emails | Varenicline + Motivational Emails
Started | 258 | 365 | 264
Completed | 185 | 137 | 165
Not Completed | 73 | 228 | 99
Not completed — Lost to Follow-up | 73 | 228 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion + Motivational Emails | Motivational Emails | Varenicline + Motivational Emails | Total
Number analyzed (Participants) | 258 | 365 | 264 | 887
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.2) | 38.6 (12.0) | 44.0 (12.8) | 41.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 196 | 157 | 503
  Male | 108 | 169 | 107 | 384
Region of Enrollment [Number; unit: participants]
  Canada | 258 | 365 | 264 | 887
Education level- less than high school diploma [Count of Participants; unit: Participants] — Number of participants with less than high school diploma
  Participants | 59 | 94 | 58 | 211
Annual household income:$20,000 or less [Count of Participants; unit: Participants] — number participants with annual income equal or less than $20,000
  Participants | 116 | 164 | 93 | 373
# Participants currently employed [Count of Participants; unit: Participants] — Number of participants who report being employed
  Participants | 136 | 198 | 138 | 472
# cigarettes smoked per day [Number; unit: participants] — # participants in cpd smoking category
  participants
    10-19 cpd | 81 | 131 | 87 | 299
    20-29 cpd | 133 | 186 | 138 | 457
    30 + cpd | 44 | 48 | 39 | 131
# participants who smoke first morning cigarette within 5 minutes [Count of Participants; unit: Participants] — # participants who report smoking first morning cigarette within 5 minutes after waking-up.
  Participants | 122 | 186 | 118 | 426
Years since started smoking daily [Mean (Standard Deviation); unit: years] — Mean (SD) years since started smoking daily
  years | 29.7 (12.1) | 24.2 (12.0) | 30.0 (12.7) | 27.5 (12.2)
# participants with less than 3 quit attempts [Count of Participants; unit: Participants] | 140 | 220 | 118 | 478
Confidence in Quitting [Mean (Standard Deviation); unit: units on a scale] — 10 point scale from: 1- Very little confidence quitting ...to.. 10-Very confident in quitting
  units on a scale | 7.8 (2.2) | 7.5 (2.1) | 7.8 (2.0) | 7.7 (2.1)
# Participants who report previous use of smoking cessation medication [Count of Participants; unit: Participants] — # participants who report previous use of medication for smoking cessation
  Participants | 142 | 186 | 142 | 470
# participants with longest period of abstinence from smoking- less than 1 week [Count of Participants; unit: Participants] — # participants who report longest period of abstinence from smoking of less than 1 week
  Participants
    less than 1 week | 75 | 115 | 74 | 264
    1 week or more | 183 | 250 | 190 | 623
Participants who report all or most of my friends smoke [Count of Participants; unit: Participants] — self report: Proportion of friends that smoke - all or most of my friends smoke
  Participants | 80 | 180 | 84 | 344
Lives with other smoker(s) [Count of Participants; unit: Participants] — Yes- lives with other smokers
  Participants | 140 | 219 | 139 | 498
History of drug or alcohol problem [Count of Participants; unit: Participants] — Self report history of alcohol or drug problem
  Participants | 40 | 55 | 27 | 122

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence of Abstinence
Description: 7-day point prevalence of abstinence was assessed by the question "Have you had a cigarette, even a puff, in the past 7 days?"
Time Frame: 6-month
Population: Number of eligible participants who either received bupropion + motivational emails, varenicline + motivational emails or motivational emails alone (because they either did not attend a physician visit or their physician decided not to prescribe them bupropion or varenicline)
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion + Motivational Emails | Motivational Emails | Varenicline + Motivational Emails
Number analyzed (Participants) | 185 | 137 | 165
Participants | 45 | 22 | 50

2. Primary Outcome: Proportion of Eligible Participants Who Were Able to Attend an Appointment With a Physician
Description: Proportion of eligible participants who were able to attend an appointment with a physician to have the prescription signed
Time Frame: End of Treatment
Population: total number of eligible participants in study
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Participants: All participants who were eligible to receive medication
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 893
Participants | 588

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Bupropion + Motivational Emails | Motivational Emails | Varenicline + Motivational Emails
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes